CLINICAL TRIAL: NCT06300957
Title: Help Wanted: Evaluating a Prevention Intervention for People With Sexual Interest in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Barry University (Other); University of Massachusetts, Lowell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00023124; CE003310 (Other Grant/Funding Number: CDC); OMB NO: 0920-1301 (Other: OMB)
Record Dates: First submitted 2024-02-22; First posted 2024-03-08 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Program Evaluation; Child Sexual Abuse; Perpetration of Child Sexual Abuse; Prevention Intervention

STUDY DESIGN:
Intervention Model Description: In Phase one investigators will recruit 10 participants to test out the study protocols. All 10 participants will go through the same study procedures.
  In Phase two, investigators will recruit 300 participants to take part in the RCT, 200 in the HW group and 100 in the WL group. After consenting to participate and completing the first online survey, participants will be randomized to either an intervention condition (N =200) or wait-list control condition (N =100) using a 2:1 allocation. The intervention group will gain access to Help Wanted for 1 month after which the participants will complete a post-intervention survey and then a three-month follow up survey. Participants in the control group will receive alternative resources for one month, then complete a one-month post-waitlist survey before being granted access to Help Wanted for a one-month period. The control group participants will then complete a one-month post-intervention survey and three-month follow-up survey.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be randomly assigned 2:1 to Experimental or Waitlist Control conditions. Experimental group will immediately access "Help Wanted", a secondary prevention program for adults who self-identify as having sexual attraction to children. Help Wanted is an online self-help curriculum to prevent Child Sexual Abuse (CSA) and reduce the psychosocial stressors of help-seekers. Content is designed to increase knowledge about CSA, counter distorted attitudes and cognitions, cope with sexual thoughts and urges about children, support development of a healthy sexuality, counter stigma and shame, build a positive self-image, and encourage safe disclosure practices. Harm and risks are clearly identified within an overall positive messaging framework. Help Wanted incorporates testimonials from survivors and from positive role models, avoids the collection of personal identifiers or reportable information, and adheres to other best practices of prevention programming.
  Interventions: Other: Help Wanted Prevention Intervention
- Waitlist Control (Other): Participants randomized to the Waitlist Control group will be barred from accessing the Help Wanted program for a period of one month.
  Interventions: Other: Waitlist Control

INTERVENTIONS:
Other: Help Wanted Prevention Intervention — The intervention includes an introductory welcome place, five training sessions that deliver core intervention content, and a resources page that provides links to external sources of support.
  The Help Wanted Prevention Intervention is a free, online, self-help course to address the needs of people with a sexual attraction to children. Help Wanted aims to provide knowledge, skills, and resources to support help-seekers' commitments to living safe, healthy, and fulfilling lives.
  Arms: Intervention
Other: Waitlist Control — Participants will be provided with information on how to access alternative resources and help lines to support mental health, suicide prevention, and child sexual abuse prevention. After one month, they will be granted access to Help Wanted.
  Arms: Waitlist Control

SUMMARY:
This project aims to evaluate the Help Wanted Prevention Intervention, an online program to provide people with a sexual attraction to children the skills and resources to support their commitment to keep children safe and to improve the participants well-being. In phase one, ten men with a sexual attraction to children who have never had a contact offense with a child will be asked to go through an abbreviated version of the participant procedures that will be used in study phase two (described next). Specifically, the ten participants will complete one of the online surveys, review the Help Wanted program, and participate in a 30-60 minute anonymous audio call with a member of the study team to provide feedback on the study procedures and materials (e.g., consent form, recruitment form). Feedback from phase one will inform changes to study procedures for phase two. Phase two consists of a large-scale evaluation of the Help Wanted program. Three hundred men with a sexual attraction to children who have never had a contact offense with a child or accessed the Help Wanted Program will be randomly selected to be part of one of two groups: the program group (N = 200) or the control group (N = 100). Both groups will be asked to complete an online survey before reviewing the Help Wanted Program, provide feedback on the program over a one-month period, and complete another online survey immediately after reviewing the program and three months after reviewing the program. Participants in the control group will have a one month waiting period after the first online survey, during which the participants will receive alternative resources and supports for mental health and sexual attraction to children. After the one month waiting period, participants in the control group will complete one additional online survey before reviewing the Help Wanted program and completing the two final online surveys (one immediately after reviewing the program, one three months after reviewing the program). Survey questions will ask about participants thoughts, feelings, and behaviors, including questions about the participants overall well-being and sexual attraction to children. All study materials and resources are in English. Resources provided to participants are also in English, but provide services in over 30 countries to include participants who may reside in countries outside of the United States. Participation is anonymous and all data will be kept confidential.

DETAILED DESCRIPTION:
The study seeks to conduct a randomized controlled trial (RCT) to evaluate the Help Wanted Prevention Intervention (Help Wanted). Help Wanted is a novel, online, self-paced intervention designed to support the needs of people with a sexual attraction to children, who wish to keep children and themselves safe. The intervention includes an introductory welcome place, five training sessions that deliver core intervention content, and a resources page that provides links to external sources of support.

The RCT will be conducted in two phases to a) evaluate the effects of Help Wanted on child sexual abuse offense behaviors, grooming behaviors, and proclivity to offend, as well as the impact on targeted psychosocial stressors that are associated with child sexual abuse perpetration; and b) examine psychosocial stressors both as outcome measures and as potential mediators and moderators.

In phase one, the investigators will beta-test RCT study procedures with a sample of adults with a sexual attraction to children who have never abused a child (N = 10). Participants in this phase will be asked to:

1. Provide a non-identifying email address to receive correspondence from the study team and verify the correspondence is working (i.e., reminders to complete assessments, a link to access study surveys and Help Wanted)..
2. Complete the pre-intervention survey (approximately 20-30 minutes).
3. Complete (i.e., click through) each of the five Help Wanted sessions and review the resources page.
4. Complete the post-intervention survey (approximately 20-30 minutes).
5. Participate in a 30-60-minute anonymous audio call (e.g., Zoom) with a member of the study team to discuss their feedback on the study procedures. These calls will be scheduled between the participant and a study staff using the participant's non-identifying email address and will take place over an online platform such as Zoom that allows participants to take part in an audio-only meeting by only providing their non-identifying email address. When using an online audio call platform, anonymity of participants will be protected by disabling video and no personal identifiable information will be collected during the call. Calls will be audio-recorded and transcribed to ensure that concerns are accurately captured and addressed as needed.

The pre-intervention and post-intervention surveys contain all survey measures so the investigators will not require beta participants to complete the additional survey (i.e., the 1-month post-intervention survey), which includes only a portion of the measures in the pre- and post-intervention surveys. Information gathered from beta participants will only inform changes to the study procedures before launching phase two of the RCT.

In phase two, the investigators will conduct a RCT to evaluate Help Wanted. Three hundred men with a sexual attraction to children who have never harmed a child will be randomly assigned to the Help Wanted intervention condition (HW; n = 200) or to a 1-month waitlist condition (WL; n = 100). HW participants will be assessed at three timepoints: recruitment (baseline), after reviewing the HW intervention for 1-month (post-intervention), and at 3-months post-intervention (follow-up). WL participants will be assessed at recruitment (baseline), after being provided alternative resources as a control for 1-month (2nd baseline), after reviewing the HW intervention for 1 month (post-intervention), and at 3-months post-intervention (follow-up). Thus, the RCT broadly follows a 2 (interventions) x 2 (timepoints) factorial design.

The alternative resources provided to the waitlist control group will include suicide prevention, mental health, and CSA prevention helplines. Specific resources for Australia, Canada, the United Kingdom, and the US, as well as a link to a list of suicide prevention, mental health, and emergency contact numbers in over 30 countries to provide additional resources for English speaking participants who may reside in these areas.

Data include measures of offense-related outcomes, internalizing problems, social deficits, sexual problems, offense-supportive cognitions, externalizing problems, adverse childhood experiences, as well as demographics.

Recruitment: The study team will design communications and plans to promote the study recruitment flyers for the beta test and RCT samples. Recruitment flyers will be provided to organizations and people who provide resources and support for people with a sexual attraction to children. These organizations will assist in recruitment by sharing the study recruitment flyer with people who utilize their services and, for the RCT, with others who may know people that may be eligible to participate in the study.

Screening Procedures: In order to monitor the number of participants in the study and ensure all study participants (in each phase) meet eligibility criteria, study team members will manually screen participants using an audio only call before allowing the participants to enroll in the study. Using approaches from a previous study with this population, all interested people will be asked to fill out a scheduling form with a date/time the participants are available to speak to a study team member and a non-identifying email address that can be used to confirm the screening call and provide the potential participant with the audio call information. Using a non-identifying email address will allow participants to remain anonymous throughout all study activities. A link with instructions on how to create a non-identifying email address will be provided on the recruitment form and the scheduling page. The scheduling form will also provide a link to a Portable Document Format (PDF) version of the appropriate Institutional Review Board-approved consent form so the participants are aware of the study details before scheduling a screening call. When an interested person signs up for a time, the participants will receive an email to their non-identifying email address with a Zoom link to complete the audio call. A trained study team member will conduct these screening calls and any responses that are not easily determined as eligible or ineligible will be run by a study investigator for review before the interested person is invited to proceed to the consent stage of the study. Screening calls are anticipated to last about 5 minutes. People who do not respond to an asked question or are deemed to not meet the study eligibility criteria will not be enrolled in the study. Ineligible people will be provided with a set of resources for general mental health, suicide prevention, and CSA prevention to the email address the participant provided. People who meet eligibility requirements will be provided with a secure study link to access the online consent form, which will be housed within the Quest system, a data collections platform.

People who are deemed eligible to participate based on their responses to the study screening questions, will be provided with a secure study link to access an Institutional Review Board (IRB) approved consent document through the Quest system (a data collections platform). The secure study link will be provided by the recruitment team via an email to the non-identifying email address the potential participant provided. Upon logging in to Quest, each participant will be required to complete a consent form before participating in any study activities. Consent documents will not ask for any identifying information (e.g., name, date of birth) and both the screening questions and consent form will only ask for information to confirm the person is eligible to participate in the study (e.g., age). People who consent yes will automatically be provided with access to the baseline survey (within Quest) to begin participation in the study.

RCT Data Analysis: the investigators will assess the pre-post effects of Help Wanted on primary outcomes (i.e., offense behaviors, and proclivity to offend) and targeted psychosocial stressors (e.g., cognitions/attitudes, coping skills, self-image) using analysis of covariance.

In an analysis of covariance (ANCOVA) study in which means of the two groups with 2:1 allocation is to be compared; the investigators estimated a total sample size of 150-300 to detect an effect size of 0.30-0.10. The total sample of 150-300 subjects achieves 80-90% power to detect differences among the means versus the alternative of equal means using an F test with a 0.05 significance level. A target sample size of 300 participants should suffice if the investigators assume a dropout rate of 15%.

The investigators will also conduct a series of mediation and moderation analyses. The mediation analyses will examine the potential mediating role of change in secondary outcomes (i.e., psychosocial stressors in five dynamic risk domains) in the association between change in primary outcomes and intervention status (HW vs. WL). The estimated sample size of 300 in Aim 1 will have 90-100% power to detect a mediation effect of at least 0.40 (regression coefficient of the mediator variable).

To test for moderation the investigators will assess whether Adverse Childhood Experiences (ACE), a pre-randomization characteristic uncorrelated with the intervention condition, moderates or buffers the association between change in primary outcomes and intervention status (i.e. intervention outcome is conditional on the level of ACEs experienced).

Data management: The security and confidentiality of data is of the utmost concern and appropriate data management procedures have been established to ensure confidentiality. The confidential nature of the data will be maintained by using study identifiers(SID)s. A limited number of study staff will have access to a linking document containing the only possible identifying information for participants, the participants non-identifying email address. This linking document will be destroyed once all data have been collected, downloaded from the Quest system (described below), cleaned, and analyzed.

Data will be collected using Quest, a data collection program. Participants will access Quest using the participants non-identifying email address and a password the participants create. All study data will be collected anonymously; therefore, no data will be connected to participant personal information. The confidentiality and security of data files on staff computers will be maintained by ensuring password protection on all computer accounts and storage of all data on Johns Hopkins University (JHU) One Drive. Electronic backup of all database files will occur daily per JHU backup procedures. Access to all study forms will be password protected and available only to the study team.

The use of an online consent form will allow participants to retain anonymity. All audio data (from phase 1 interviews) will be encrypted and saved on JHU One Drive until it is transcribed and analyzed, at which point audio files will be permanently destroyed. Access to all data will be password protected and data will be backed up daily to a secure location on the Quest system (for phase one and two survey data) and on JHU One Drive (for phase one audio data and linking document).

Any study problems or concerns will be brought to the attention of the project manager and PI immediately and the IRB and Centers for Disease Control will be notified according to IRB policies (when applicable). Three experts selected for the ability to comprehend clinical research data, understanding of the population under study, or understanding of prevention interventions were selected to serve on a Data Safety Monitoring Board (DSMB) for this project. The DSMB will meet bi-annually throughout the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Men (cis-gender and transgender)
* Age 18 and older (no upper age limit)
* Self-identified sexual attraction to prepubescent or early pubescent children
* No prior contact offense with a child
* Never accessed the Help Wanted intervention.

Exclusion Criteria:

* Women (cis-gender and transgender)
* Under age 18
* No sexual attraction to prepubescent or early pubescent children
* Any prior contact offense with a child
* Previously accessed the Help Wanted intervention

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cisgender and transgender men are eligible
Enrollment: 310 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Sexual Behavior Involving Minors Scale (SBIMS). | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  8 items; score range from 8 to 40; higher scores indicate more problem behavior.
Sexual Child Molestation Risk Assessment (SChiMRA) score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  6 items; scores involve marking an X on a slide rule from "very likely" to "not at all likely or nearly every day"; marks further to the right indicate higher risk.

SECONDARY OUTCOMES:
Depression, Anxiety and Stress Scale-21 (DASS-21) | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  21 items; score range from 0 to 63; higher scores indicate worse severity.
Suicidal Ideation Attributes Scale (SIDAS) | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  5 items; score range from 0 to 50; higher score indicates higher suicidal ideation.
General Self-Efficacy Scale - Short Form (GSE-6). | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  6 items; score range from 6 to 24; higher scores indicate greater self-efficacy.
Revised University of California, Los Angeles (UCLA) Loneliness Scale | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  10 items; score range from 10 to 40; higher scores indicate more loneliness.
Self-Efficacy Scale Related to Minors (SESM) | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  30 items; score range from 30 to 120; higher scores indicate greater self-efficacy.
Hypersexual Behavior Inventory-19 score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  19 items; score range from 19 to 95; higher scores indicate higher levels of sexual thoughts.
Sexual Attraction to Children | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  14 items; responses are descriptive only.
Cognitions of internet sexual offending score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  28 items; score range from 28-112; higher scores indicate more support for offending.
Cognitions that condone and support sexual offending against children scale - short form | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  10 items; score range from 10-40; higher scores indicate more offense supportive cognitions.
Emotional Congruence with Children score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  12-items; score range from 12-48; higher scores indicate more congruence.
Brief Aggression Questionnaire score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  12-items; score range from 12-60; higher scores indicate more aggression.
Short Self-Regulation Questionnaire score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  31 items; score range from 31-155; higher scores indicate greater self-regulation
Alcohol Use Disorders Identification Test (AUDIT) score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  10 items screen for problematic alcohol use; score range from 0-40; higher scores indicate greater use.
Recent Alcohol & Cannabis Use score | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  2 items; each scored 1-7; higher score indicates more frequent use.

OTHER OUTCOMES:
Demographic characteristics as assessed by survey developed by study team | Baseline
  15 items; responses are descriptive only.
Number of Sexual Health Services Used | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  9 items; responses are descriptive only.
Sexual Offence Self-Report Risk Scale (SOSRS): | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  6 items; responses are descriptive only.
Minor Attraction Outness Scale | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  11-items; responses are descriptive only.
Revised Adverse Childhood Experiences Scale | Baseline
  14 items; responses are descriptive only.
Balanced Inventory of Desirable Responding - Impression Management Subscale (BIDR-Version 6-Form 40 - IMS). | Baseline
  16 items; score range from 16-112; higher scores indicate more desirable responding.
Impact of Research Participation as assessed by survey | Baseline, 1 month post waitlist (waitlist only), 1 month post-intervention, 3 months
  Closing Questions: Assessing the Impact of Research Participation. 7 items; each item has a distinct response option (e.g., open-text; sliding scale; likert-type scale).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth J Letourneau, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shields RT, Murray SM, Ruzicka AE, Buckman C, Kahn G, Benelmouffok A, Letourneau EJ. Help wanted: Lessons on prevention from young adults with a sexual interest in prepubescent children. Child Abuse Negl. 2020 Jul;105:104416. doi: 10.1016/j.chiabu.2020.104416. Epub 2020 Feb 17. PMID 32081437
- See also: Help Wanted is an online, self-paced intervention designed to support the needs of people with a sexual attraction to children, who wish to keep children and themselves safe. — http://helpwantedprevention.org